CLINICAL TRIAL: NCT05076279
Title: Safety and Efficacy of Single or Reduced Ports Laparoscopic Gastrectomy for Advanced Gastric Cancer (SPACE-01) Phase II Clinical Trial
Brief Title: Safety and Efficacy of Single or Reduced Ports Laparoscopic Gastrectomy for Advanced Gastric Cancer (SPACE-01)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yun-Suhk Suh, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-2107-696-001
Record Dates: First submitted 2021-09-29; First posted 2021-10-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma
Keywords: Gastric cancer; Gastric adenocarcinoma; Gastrectomy; Single port
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single port or reduced ports (Experimental): Single port or reduced ports laparoscopic distal gastrectomy and D2 lymph node dissection
  Interventions: Procedure: Single port or reduced ports laparoscopic distal gastrectomy and D2 lymph node dissection

INTERVENTIONS:
Procedure: Single port or reduced ports laparoscopic distal gastrectomy and D2 lymph node dissection — Single port or reduced ports laparoscopic distal gastrectomy and D2 lymph node dissection

SUMMARY:
The aim of this study is to verify the safety and efficacy of single or reduced ports laparoscopic gastrectomy for advanced gastric cancer.

DETAILED DESCRIPTION:
Since two cases of single-incision laparoscopic gastrectomy in early gastric cancer were reported in 2011, the safety and efficacy of single-incision laparoscopic gastrectomy in early gastric cancer have been reported several times.

Recently, the feasibility of laparoscopic single-incision gastrectomy in some advanced gastric cancer has already been reported.

The total number of retrieved lymph nodes during gastric cancer surgery is one of the most important indicators for securing oncological safety and predicting the therapeutic effect in gastric cancer surgery.

Therefore, in order to prospectively evaluate the efficacy of single-incision or reduced-port laparoscopic gastrectomy for advanced gastric cancer as an oncological operation, the purpose of this study is to evaluate the number of resected lymph nodes after D2 lymph node dissection in single-incision or reduced-port laparoscopic gastrectomy for advanced gastric cancer.

All surgeries are performed as single-incision laparoscopic surgery using a 3-4 cm umbilical incision, and D2 lymph node dissection is performed according to the Japanese gastric cancer treatment guidelines 2018 by the Japanese Gastric Cancer Association.

When an additional trocar is required, it is classified as reduced port laparoscopy when one additional trocar is added.

For surgical assistance, including effective visual field development during surgery, a self intra-corporeal retractor (FJ clip®, or Internal organ retractor®) or an additional trocar (up to 1 trocar) could be used.

An articulating laparoscopic surgical instrument (Artisential ®) can be used for safe access to difficult areas of the D2 lymph node dissection, such as the superior border of the pancreas.

Before the end of the surgery, the surgeon evaluates the completeness of D2 lymph node dissection and radical resection of the primary tumor(R0 resection). If insufficient, the operation is converted to multi-port laparoscopic surgery or open surgery, and additional D2 lymph node dissection and tumor resection are performed, and those cases are recorded separately in the registry as multiport/open conversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have confirmed that participants have advanced gastric cancer at clinical stage T2 or higher and who can undergo distal gastrectomy for primary gastric cancer who have consented to single-port and reduced-port laparoscopic gastric cancer surgery
* Patients diagnosed with locally advanced gastric cancer in which no enlarged lymph nodes were observed in the preoperative examination, or lymph node metastases confined to the left gastric artery or perigastric area were suspected.
* Those who have not been treated for systemic inflammatory disease before surgery

Exclusion Criteria:

* Those who have previously had gastrectomy.
* Those who have a laparotomy except for appendectomy, cholecystectomy or cesarean section.
* Patients with clinical (preoperative or intraoperative) stage T4b accompanied by infiltration of surrounding organs
* Those with bulky lymph nodes (single nodules over 3 cm or multiple nodules over 1.5 cm)
* Patients with confirmed distant metastasis (M1)
* Severe liver cirrhosis
* Patients who is judged by the investigator to be inappropriate for this study
* Patients who are taking antithrombotic drugs, including antiplatelet drugs and anticoagulants, and cannot safely stop before surgery

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
number of retrieved lymph nodes | during operation
  number of retrieved lymph nodes during operation

SECONDARY OUTCOMES:
postoperative complications | 3 year
  Postoperative complications are problems that can happen after participants have had surgery but which were not intended.
Quality of life of the participants | before surgery (within 1 month before the day of surgery), within 1 week after surgery, within 1 month after surgery, within 3 months after surgery, within 6 months after surgery, and within 12 months after surgery
  The patient's quality of life is assessed using the widely used quality of life questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), sto22) before surgery (within 1 month before the day of surgery), within 1 week after surgery, within 1 month after surgery, within 3 months after surgery, within 6 months after surgery, and within 12 months after surgery, respectively.
3 year relapse-free survival | 3 year
  3 year relapse-free survival

CONTACTS AND LOCATIONS:
Overall Officials: YunSuhk Suh, M.D., Ph.D., Principal Investigator — ysksuh@gmail.com
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JH, Lee MS, Kim HH, Park DJ, Lee HJ, Yang HK, Park KU. Comparison of single-incision laparoscopic distal gastrectomy and laparoscopic distal gastrectomy for gastric cancer in a porcine model. J Laparoendosc Adv Surg Tech A. 2011 Dec;21(10):935-40. doi: 10.1089/lap.2011.0280. Epub 2011 Nov 1. PMID 22044252
- [Background] Omori T, Fujiwara Y, Moon J, Sugimura K, Miyata H, Masuzawa T, Kishi K, Miyoshi N, Tomokuni A, Akita H, Takahashi H, Kobayashi S, Yasui M, Ohue M, Yano M, Sakon M. Comparison of Single-Incision and Conventional Multi-Port Laparoscopic Distal Gastrectomy with D2 Lymph Node Dissection for Gastric Cancer: A Propensity Score-Matched Analysis. Ann Surg Oncol. 2016 Dec;23(Suppl 5):817-824. doi: 10.1245/s10434-016-5485-8. Epub 2016 Aug 10. PMID 27510844
- [Background] Omori T, Fujiwara Y, Yamamoto K, Yanagimoto Y, Sugimura K, Masuzawa T, Kishi K, Takahashi H, Yasui M, Miyata H, Ohue M, Yano M, Sakon M. The Safety and Feasibility of Single-Port Laparoscopic Gastrectomy for Advanced Gastric Cancer. J Gastrointest Surg. 2019 Jul;23(7):1329-1339. doi: 10.1007/s11605-018-3937-0. Epub 2018 Sep 5. PMID 30187335